CLINICAL TRIAL: NCT06378294
Title: Locoregional Control With Radiotherapy of cT1-2N0 Invasive Breast Cancer Patients With MACrometastases in the Sentinel Node Treated With MAstectomy: a Multi-center Observational Study
Brief Title: Locoregional Control With Radiotherapy of Breast Cancer Patients With MACrometastases Treated With MAstectomy (MACMA)
Acronym: MACMA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital A Coruña (Other)
Collaborators: Complejo Hospitalario Universitario de Pontevedra (Other); Complejo Hospitalario Universitario de Vigo (Other); Complejo Hospitalario Universitario de Santiago (Other); Hospital Universitario Lucus Augusti (Other); Complexo Hospitalario de Ourense (Other); Hospital Arquitecto Marcide (Other)
Responsible Party: Principal Investigator, Alberto Bouzon, Principal Investigator, M.D., Ph.D., University Hospital A Coruña
Other Study IDs: UHACoruna
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: axillary radiotherapy; mastectomy; sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mastectomy patients: clinically node-negative T1-2 invasive breast cancer patients treated with upfront mastectomy
  Interventions: Procedure: Mastectomy

INTERVENTIONS:
Procedure: Mastectomy — Adjuvant postmastectomy radiotherapy
  Other Names: Axillary radiotherapy without axillary lymph node dissection

SUMMARY:
Sentinel lymph node biopsy (SLNB) is the standard procedure to stage the axilla in clinically node-negative invasive breast cancer (IBC) patients undergoing upfront surgery.

The ACOSOG-Z0011 and the AMAROS trial demonstrated that SLNB with or without radiotherapy provided equivalent local control and survival to axillary lymph node dissection (ALND) in early-stage breast cancer patients with 1 or 2 positive SLNs. However, the ACOSOG-Z0011 trial did not included patients treated with mastectomy, and the AMAROS trial only included 17% of mastectomy patients.

The investigators conduct an observational cohort study of early stage breast cancer patients receiving upfront mastectomy with 1 or 2 macrometastases after SLNB. The study aim to demonstrate a 5-year disease-free survival of not less than 80% when ALND is omitted and replaced by axillary radiotherapy, and determine the axillary recurrence rate.

DETAILED DESCRIPTION:
This is a multi-center, prospective study with an estimated sample size of 60 early-stage IBC patients.

Clinically node-negative T1-2 IBC patients undergoing mastectomy with up to 2 macrometases after SLNB will be informed about this study.

Patients will be checked with annual mammography and clinical examination. The axilla will be checked with ultrasound at 3 and 5 years of the surgery.

After surgery, patients will receive axillary radiotherapy, but no ALND, and adjuvant systemic treatment based on international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T1-2 primary invasive breast cancer
* No suspicion of lymph node involvement prior to sentinel lymph node biopsy
* Patients undergoing upfront mastectomy
* Macrometastasis in not more than 2 lymph nodes at sentinel lymph node biopsy
* Patients treated with adjuvant axillary radiotherapy

Exclusion Criteria:

* Prior history of invasive breast cancer
* Medical contraindication for radiotherapy
* Medical contraindication for adjuvant systemic treatment
* Planned neoadjuvant systemic treatment
* Distant metastasis at initial diagnosis
* Inability to absorb or understand the meaning of the study information

Ages: 18 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Early-stage invasive breast cancer patients receiving upfront mastectomy
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 and 5 years
  recurrence in the ipsilateral breast/thoracic wall, regional recurrence, distant recurrence or death
Axillary recurrence rate | 3 and 5 years
  recurrence rate in the ipsilateral axillary lymph nodes

SECONDARY OUTCOMES:
Overall survival | 5 years
  any cause of death as event

CONTACTS AND LOCATIONS:
Overall Officials: ALBERTO BOUZÓN, Principal Investigator — HOSPITAL UNIVERSITARIO A CORUÑA
Locations (7):
- Spain (7):
  - Hospital Universitario Ferrol, Ferrol, A Coruña
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital Universitario Vigo, Vigo, Pontevedra
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Lugo, Lugo
  - Hospital Universitario Ourense, Ourense
  - Hospital Universitario Pontevedra, Pontevedra

IPD SHARING:
Plan to Share IPD: No
Results will be published by the investigators in academic journals

REFERENCES:
- [Result] Giuliano AE, Ballman KV, McCall L, Beitsch PD, Brennan MB, Kelemen PR, Ollila DW, Hansen NM, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, Hunt KK, Morrow M. Effect of Axillary Dissection vs No Axillary Dissection on 10-Year Overall Survival Among Women With Invasive Breast Cancer and Sentinel Node Metastasis: The ACOSOG Z0011 (Alliance) Randomized Clinical Trial. JAMA. 2017 Sep 12;318(10):918-926. doi: 10.1001/jama.2017.11470. PMID 28898379
- [Result] Bartels SAL, Donker M, Poncet C, Sauve N, Straver ME, van de Velde CJH, Mansel RE, Blanken C, Orzalesi L, Klinkenbijl JHG, van der Mijle HCJ, Nieuwenhuijzen GAP, Veltkamp SC, van Dalen T, Marinelli A, Rijna H, Snoj M, Bundred NJ, Merkus JWS, Belkacemi Y, Petignat P, Schinagl DAX, Coens C, van Tienhoven G, van Duijnhoven F, Rutgers EJT. Radiotherapy or Surgery of the Axilla After a Positive Sentinel Node in Breast Cancer: 10-Year Results of the Randomized Controlled EORTC 10981-22023 AMAROS Trial. J Clin Oncol. 2023 Apr 20;41(12):2159-2165. doi: 10.1200/JCO.22.01565. Epub 2022 Nov 16. PMID 36383926